CLINICAL TRIAL: NCT05410262
Title: Specific Mechanical Power Assessment in Patients With Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Nestor Pistillo, Head of Intensive Care Unit al Hospital El Cruce, Hospital El Cruce
Other Study IDs: El Cruce
Record Dates: First submitted 2022-06-01; First posted 2022-06-08 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Ventilation, Mechanical
Keywords: ARDS; Mechanical power
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanical power and risk of ventilator-induced lung injury in patients with ARDS: This study will prospectively evaluate patients consecutively admitted with ARDS, as defined according to the Berlin expert consensus
  Interventions: Other: Evaluation of CT images

INTERVENTIONS:
Other: Evaluation of CT images — A helicoidal CT scanner will be used (Aquilion CXL, Toshiba, Japan), with AIDR 3D technique (Adaptive Iterative Dose Reduction 3D) in order to minimize exposure to X-rays. Two complete thorax CT scans will be performed, one of them in expiratory pause (PEEP) and the other in inspiratory pause (PPlat). Esophageal pressure shall be measured (FluxMed GrT, Argentina) and transpulmonary pressure will be calculated at the end of inspiration (Ppl-insp) and expiration (Ppl-exp).
  Other Names: Evaluation of transpulmonary pressures

SUMMARY:
In ARDS patients, mechanical ventilation should minimize ventilator-induced lung injury. The mechanical power which is the energy per unit time released to the respiratory system according to the applied tidal volume, PEEP, respiratory rate, and flow should reflect the ventilator-induced lung injury

DETAILED DESCRIPTION:
Mechanical ventilation is an essential tool for the treatment of patients with acute respiratory distress syndrome (ARDS); however, as other strategies, it is not free of complications. Inadequate ventilation may have a negative impact on the lung that may eventually cause the development of multiple organ failure and death. This process is known as ventilator-induced lung injury (VILI). From a clinical perspective, one of the most important objectives of ARDS treatment is to avoid or mitigate the development of VILI, not only to preserve pulmonary integrity, but also to reduce mortality.

Ventilator-induced lung injury results from the interaction between the mechanical load applied to the lung and its capacity to tolerate it. Factors such as tidal volume (Vt), plateau pressure (PPlat), lung strain or insufflation pressure (ΔP), inspiratory flow rate (VI), respiratory rate (RR), excessive inspiratory effort, high levels of FiO2 and high levels of positive end-expiratory pressure (PEEP), have been directly involved in damage mechanism. With an integrating and rheological idea, the concept of mechanical power tries to encompass the majority of these factors within a measurable unit in joules per minute, as the expression of power applied on a repetitive basis on the respiratory system in ARDS. Although the concept of MP holds promise for preventing the risk of VILI, its utility has not been proven in clinical practice until now. The main value of MP over the rest of commonly used variables for the monitoring of patients with ARDS is that it includes flow on injury mechanism (kinetic energy), accepting that an inverse relationship exists between this mechanism and the capacity of alveoli to adapt to change during the ventilation cycle (strain rate), as well as it embodies the concept of process repeatability (respiratory rate), though not of its duration. This begs the question whether we should consider its value at the moment of defining a mechanical ventilation strategy. The main disadvantage of its application is that MP conceives the respiratory system in an integrated manner and not related to or standardized with the ventilable lung portion, that is ultimately the one who has to withstand the ventilatory load; in other words, the same MP may have different consequences depending on the baby lung size or its equivalent, the severity of ARDS.

The objective of this study is to evaluate the influence of the ventilable lung size on VILI mechanisms in patients suffering from ARDS treated with protective ventilation with similar MP.

ELIGIBILITY:
Inclusion Criteria: patients consecutively admitted with ARDS -

Exclusion Criteria: Patients who meet any of the following criteria: history of emphysema, asthma, pneumothorax or bronchopleural fistula. Severe instability condition at the time of the study: SaO2 ≤90%, shock requiring noradrenaline ≥0,5 γ/kg/min, ventricular arrhythmia, myocardial ischemia and endocranial hypertension. Esophageal pathology that contraindicates esophageal balloon placement. Severe coagulopathy (platelet count <20000/mm3 or INR >4). Inability to undergo CT imaging: morbid obesity (≥170 kg) or abdominal girth >200 cm. Patients with do-not-resuscitate (DNR) orders, pregnant women and those who participated in other research studies within the last 30 days.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients consecutively admitted with ARDS, as defined according to the Berlin expert consensus
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
specific mechanical power | "immediately after the intervention/procedure/surgery"
  Specific mechanical power was calculated as the ratio of mechanical power to ventilable lung volume.
relationship between lung load and severity of ARDS | "immediately after the intervention/procedure/surgery"
  relationship between specific mechanical power and severity of ARDS
relationship between lung load and elastance of ARDS | "immediately after the intervention/procedure/surgery"
  relationship between specific mechanical power and elastance of ARDS
relationship between lung load and strain | "immediately after the intervention/procedure/surgery"
  relationship between specific mechanical power and strain
relationship between lung load and atelectrauma | "immediately after the intervention/procedure/surgery"
  relationship between specific mechanical power and atelectrauma

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Pistillo, Principal Investigator — Hospital El Cruce
Locations (1):
- Hospital de Alta Complejidad en Red El Cruce Nestor C. Kirchner, San Juan Bautista, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Cressoni M, Gotti M, Chiurazzi C, Massari D, Algieri I, Amini M, Cammaroto A, Brioni M, Montaruli C, Nikolla K, Guanziroli M, Dondossola D, Gatti S, Valerio V, Vergani GL, Pugni P, Cadringher P, Gagliano N, Gattinoni L. Mechanical Power and Development of Ventilator-induced Lung Injury. Anesthesiology. 2016 May;124(5):1100-8. doi: 10.1097/ALN.0000000000001056. PMID 26872367
- [Background] Costa ELV, Slutsky AS, Brochard LJ, Brower R, Serpa-Neto A, Cavalcanti AB, Mercat A, Meade M, Morais CCA, Goligher E, Carvalho CRR, Amato MBP. Ventilatory Variables and Mechanical Power in Patients with Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2021 Aug 1;204(3):303-311. doi: 10.1164/rccm.202009-3467OC. PMID 33784486
- [Background] Coppola S, Caccioppola A, Froio S, Formenti P, De Giorgis V, Galanti V, Consonni D, Chiumello D. Effect of mechanical power on intensive care mortality in ARDS patients. Crit Care. 2020 May 24;24(1):246. doi: 10.1186/s13054-020-02963-x. PMID 32448389
- [Background] Gattinoni L, Marini JJ, Collino F, Maiolo G, Rapetti F, Tonetti T, Vasques F, Quintel M. The future of mechanical ventilation: lessons from the present and the past. Crit Care. 2017 Jul 12;21(1):183. doi: 10.1186/s13054-017-1750-x. PMID 28701178